CLINICAL TRIAL: NCT01732367
Title: Randomized Trial of Tenofovir Versus Lamivudine Plus Adefovir in Lamivudine Plus Adefovir Treated Lamivudine-resistant Chronic Hepatitis B Patients With Undetectable Hepatitis B Virus DNA.
Brief Title: TDF VS LAM + ADV in LAM + ADV Treated LAM-resistant CHB Patients With Undetectable Hepatitis B Virus DNA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Collaborators: Kyungpook National University Hospital (Other); Daegu Catholic University Medical Center (Other); DongGuk University (Other); Pusan National University Hospital (Other); Yeungnam University Hospital (Other)
Responsible Party: Principal Investigator, Jang Byoung Kuk, Keimyung University Dongsan Medical Center, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TDF0001
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Hepatitis B
Keywords: Tenofovir; Lamivudine; Adefovir; Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Lamivudine; adefovir; adefovir dipivoxil; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lamivudine plus adefovir (Active Comparator): Continue lamivudine/adefovir add on treatment (standard treatment)
  Interventions: Drug: Lamivudine plus adefovir
- Tenofovir (Experimental): Switch from lamivudine/adefovir add on treatment to tenofovir monotherapy
  Interventions: Drug: Tenofovir

INTERVENTIONS:
Drug: Lamivudine plus adefovir — Lamivudine 100mg QD for 96 weeks + Adefovir 10mg QD for 96 weeks
  Other Names: Zeffix; Hepsera
  Arms: Lamivudine plus adefovir
Drug: Tenofovir — Tenofovir 300mg QD for 96 weeks
  Other Names: Viread
  Arms: Tenofovir

SUMMARY:
This study will provide a rationale for switch from lamivudine plus adefovir to tenofovir monotherapy in Lamivudine plus Adefovir Treated Lamivudine-resistant chronic hepatitis B patients with Undetectable Hepatitis B Virus DNA

DETAILED DESCRIPTION:
Recently, in Korea, long-term medication of antiviral agents and their resulting resistance expression have been the most serious cause of failure to treat chronic hepatitis B. Exp.

In particular, the annual resistance rate to lamivudine currently widely being used in Korea amounts to about 15 to 20 percents and the rate is expected to reach 70 to 80 percent in four to five years.

The guidelines by the American Association for the Study of Liver Disease (AASLD) and the European Association for the Study of the Liver (EASL) recommend a combination therapy with adefovir or tenofovir for patients with lamivudine resistant HBV .

In Korea, however, in case of combined prescription of lamivudine and adefovir, only one of them is covered by the health insurance and therefore many patients are difficult to continue treatment due to their economic conditions.

Tenofovir that has been developed most recently and will be placed on sale sooner or later in Korea has strong antiviral effects, causes little or no emergence of resistant viruses, and is known to have lower nephrotoxicity than adefovir.

In particular, several papers reported that tenofovir has effective and sustaining antiviral effects in patients who had other antiviral agents resistant HBV as well as those who received initial treatment. This shows that patients only with lamivudine resistant HBV can be treated only with tenofovir without a combination therapy and when they have low levels of HBV DNA, treatment is relatively effective despite their resistance to adefovir.

Therefore, it is considered that tenofovir switching therapy in patients with undetectable HBV DNA after lamivudine plus adefovir combination therapy to maintain their virus response.

The results of this study will provide a rationale for switch from lamivudine plus adefovir to tenofovir monotherapy in such patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 or older
* The CHB patients (both HBeAg-positive and - negative) who have at least 6 months undetectable HBV DNA (serum HBV DNA ≤ 20 IU/mL) after lamivudine plus adefovir combination therapy.

Exclusion Criteria:

* Patients with decompensated liver disease
* Patients with HCV, HDV or HIV
* Patients with HCC
* Serum ALT > 2x ULN level
* Serum creatinine > 2.0mg/dL
* Pregnant or lactating women
* Women who have a plan for pregnancy within the three coming years
* Patients who have uncontrolled severe concomitant diseases- severe cardiovascular diseases and other infection
* Those who have no capabilities to understand and sign an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2012-11; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Percentage number of patients with virus reactivation | Week 96 while on treatment
  Percentage number of patients with virus reactivation (HBV DNA > 40 IU/mL on two consecutive samples taken 1 month apart, or persistent HBV DNA levels of 20-40 IU/mL on three consecutive 1 month interval) at Week 96 while on treatment.

SECONDARY OUTCOMES:
Virologic response | Week 96 while on treatment
  Virologic response Percentage number of patients with virus reactivation at Week 48
Antiviral resistance | Week 96 while on treatment
  Antiviral resistance percentage number of patients who developed drug resistant mutation at Week 48 and 96 while on randomized therapy.
Biochemical response | Week 96 while on treatment
  Biochemical response percentage number of patients with biochemical breakthrough at Week 48 and 96
Serologic response | Week 96 while on treatment
  Serologic response (1) HBeAg loss/seroconversion in HBeAg-positive CHB Percentage number of patients with HBeAg loss or seroconversion at Week 48 and 96.
Safety assessment | Week 96 while on treatment
  Safety assessment

CONTACTS AND LOCATIONS:
Overall Officials: Byoung Kuk Jang, M.D, Principal Investigator — Department of Internal Medicine, Keimyung University Dongsan Medical Center
Locations (1):
- Department of Internal Medicine, Keimyung University Dongsan Medical Center, Daegu, South Korea

REFERENCES:
- [Derived] Lee HJ, Kim SJ, Kweon YO, Park SY, Heo J, Woo HY, Hwang JS, Chung WJ, Lee CH, Kim BS, Suh JI, Tak WY, Jang BK. Evaluating the efficacy of switching from lamivudine plus adefovir to tenofovir disoproxil fumarate monotherapy in lamivudine-resistant stable hepatitis B patients. PLoS One. 2018 Jan 12;13(1):e0190581. doi: 10.1371/journal.pone.0190581. eCollection 2018. PMID 29329305